CLINICAL TRIAL: NCT00516386
Title: Safety Profile of Insulin Like Growth Factor-1 (IGF-I) Administration in Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Tercica (Industry)
Responsible Party: Principal Investigator, Madhusmita Misra, Associate Professor of Pediatrics, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2006P-000737
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Results first posted 2011-08-04 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-10

CONDITIONS: Anorexia Nervosa
Keywords: Adolescents; Anorexia nervosa (AN); Bone formation markers; Insulin like growth factor-1 (IGF-I)
MeSH Terms: conditions — Anorexia Nervosa | interventions — mecasermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulin like growth factor- 1 (IGF-1) (Experimental): Adolescent girls with AN meeting inclusion criteria were administered recombinant human (rh) rhIGF-1 at a dose of 35-40 mcg/k twice daily by subcutaneous injections for a 7-10 day period.
  Interventions: Drug: RhIGF-1

INTERVENTIONS:
Drug: RhIGF-1 — 35-40 mcg/k/dose twice daily SC
  Other Names: Increlex

SUMMARY:
The purpose of this study was to determine whether giving insulin like growth factor-I (IGF-I) to adolescent low weight girls is safe and whether this increases levels of bone formation markers.

DETAILED DESCRIPTION:
Adolescents with anorexia nervosa (AN) are at high risk for low bone mineral density at a time when healthy adolescents are rapidly accruing bone, with implications for peak bone mass and fracture risk in later life. They are also deficient in insulin-like growth factor I (IGF-I), the bone trophic factor made in the liver in response to growth hormone (GH), despite elevated levels GH. It is possible that deficiency of IGF-I, a hormone very important for the maintenance of skeletal integrity, may contribute to the severe osteopenia seen in AN. The physiologic effects of rhIGF-I treatment in adolescents with AN had not been studied. The goal of this proposal was to investigate the acute effects of rhIGF-I on bone metabolism in adolescent girls with AN.

Specific Aim: It was hypothesized that adolescent AN patients, being IGF-I deficient, would respond to exogenously administered rhIGF-I with elevations in biochemical indices of bone turnover. Therefore, rhIGF-I was administered to AN patients by subcutaneous injection over 10 days with concomitant measurement of indices of bone turnover, and calcium regulatory hormones.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent girls with anorexia nervosa 12-18 years old

Exclusion Criteria:

* Pregnancy or nursing
* Hematocrit < 30%, K < 3 mmol/L
* Any illness (other than anorexia nervosa) known to affect bone and mineral metabolism such as diabetes, alcoholism, untreated hypo- or hyperthyroidism, or hyperparathyroidism
* History of use of any medicine, such as corticosteroids, known to affect bone density. Subjects who were on estrogen were still eligible to participate in the study.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Primary Completion 2008-05 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhu Misra, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Misra M, McGrane J, Miller KK, Goldstein MA, Ebrahimi S, Weigel T, Klibanski A. Effects of rhIGF-1 administration on surrogate markers of bone turnover in adolescents with anorexia nervosa. Bone. 2009 Sep;45(3):493-8. doi: 10.1016/j.bone.2009.06.002. Epub 2009 Jun 10. PMID 19523548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixteen anorexia nervosa patients between the ages of 12-18 years were recruited. Patients were determined by their psychiatrists to meet criteria for AN as described in the Diagnostic and Statistical Manual of Mental Disorders (a).
Pre-assignment Details: Four subjects were not interested in the study after the screen, and two were lost to follow-up.
Groups:
- RhIGF-1: All study subjects were administered rhIGF-1 at a dose of 35-40 mcg/k/dose twice daily SC for 7-10 days.
Period: Overall Study
Arm/Group | RhIGF-1
Started | 16
Completed | 10
Not Completed | 6
Not completed — not interested in the study | 4
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | RhIGF-1
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.2 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Levels of Insulin Like Growth Factor-1 (IGF-I) Following Recombinant Human (rh) IGF-1 Administration in Girls With Anorexia Nervosa
Time Frame: Baseline and 7-10 days
Population: 16 subjects were screened for the study, and 10 completed the study. 10 were analyzed.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | RhIGF-1
Number analyzed (Participants) | 10
ng/ml | 542.9 (40.9)
Statistical Analysis 1: Comparison: RhIGF-1; We used paired t-tests to assess changes in levels of IGF-1 from baseline levels in girls with AN receiving rhIGF-1. Our hypothesis was that rhIGF-1 administration would be associated with a significant increase in IGF-1 levels; Test type: Superiority or Other; p < 0.05, Paired t-test; Mean Difference (Net) = 543, Standard Error of Mean 41

2. Secondary Outcome: Change in Levels of N-terminal Propeptide of Type 1 Procollagen (P1NP) Following rhIGF-1 Administration in Girls With Anorexia Nervosa
Time Frame: Baseline and 7-10 days
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | RhIGF-1
Number analyzed (Participants) | 10
ng/ml | 39.3 (9.3)
Statistical Analysis 1: Comparison: RhIGF-1; We used a paired t-test to determine the change in P1NP from baseline to 7-10 days following administration of rhIGF-1; Test type: Superiority or Other; p < 0.05, Paired t-test; Mean Difference (Final Values) = 39.3, Standard Error of Mean 9.3

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | RhIGF-1
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 4/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RhIGF-1 (N=16)
Hospitalization for weight gain (Metabolism and nutrition disorders) | 1 (1) — Not related to study or study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RhIGF-1 (N=16)
Headaches (General disorders) | 4 (4) — Mild to moderate- not associated with raised intracranial pressure. Moderate: 3 subjects; two resolved with Tylenol or Advil Mild: 2 subjects; 1 resolved with Advil, the other did not need meds

LIMITATIONS AND CAVEATS:
A limitation of our study is that this was not a randomized controlled trial of rhIGF-1 versus placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No